CLINICAL TRIAL: NCT05813275
Title: Phase 3 Randomized Double-Blind Placebo-Controlled 6-month Parallel-Arm Study to Compare a Fixed Dose Combination of Aroxybutynin/Atomoxetine (AD109) to Placebo in Obstructive Sleep Apnea (SynAIRgy Study)
Brief Title: Parallel-Arm Study to Compare AD109 to Placebo With Patients With OSA (SynAIRgy Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APC-APN-305
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: OSA
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AD109 (Experimental): AD109
  Interventions: Drug: AD109
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AD109 — Oral administration at bedtime
  Arms: AD109
Drug: Placebo — Oral administration at bedtime
  Arms: Placebo

SUMMARY:
This is a Phase 3 Randomized Double-Blind Placebo-Controlled 6-month Parallel-Arm Study to Compare a Fixed Dose Combination of AD109 to Placebo in Obstructive Sleep Apnea.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at the time of informed consent.
2. PSG criteria: AHI of ≥10 and ≤45; ≤ 25% central or mixed apneas; and PLM arousal index ≤15
3. PROMIS-Fatigue: raw score ≥17
4. PAP intolerance or current PAP refusal.
5. BMI between 18.5 and 40 kg/m2 for men, or 42 kg/m2 for women, inclusive.

Exclusion Criteria:

1. Narcolepsy, restless leg syndrome, REM sleep behavior disorder
2. Insomnia disorder characterized by difficulty initiating or maintaining sleep, or use within the past month of sedative-hypnotics or other medication for the purpose of treating or avoiding insomnia symptoms.
3. Pierre Robin, Treacher Collins, or other craniofacial malformation syndrome, or grade ≥3 tonsillar hypertrophy.
4. Clinically significant cardiac disease, e.g., ventricular arrhythmia, untreated or unstable coronary artery disease, cardiac failure. Stable atrial arrhythmia is allowed.
5. Neuromuscular disorder (e.g., motor neuron disease, muscular dystrophy or myopathy, myasthenic syndrome); epilepsy; Parkinson, Alzheimer, or other neurodegenerative disease.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2023-09-16 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Apnea-Hypopnea Index (AHI) | 6 months
  AHI, Apnea-Hypopnea Index, is the number of apneas or hypopneas recorded via polysomnography during the study per hour of sleep. Apnea is defined as a cessation of airflow lasting at least 10 seconds, hypopnea as a decrease in airflow by at least 30% from baseline for at least 10 seconds occurring with a drop in oxygen saturation (SpO2) by at least 4%.

CONTACTS AND LOCATIONS:
Locations (73):
- United States (65):
  - Alabama Neurology & Sleep Medicine, Tuscaloosa, Alabama
  - Desert Clinical Research - CCT Research, Mesa, Arizona
  - Foothills Research Center - CCT Research, Phoenix, Arizona
  - Fiel Family Sports Medicine - PC CCT Research, Tempe, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Orange County Research Institute, Anaheim, California
  - North County Neurology Associates, Carlsbad, California
  - Core Healthcare Group, Cerritos, California
  - Exalt Clinical Research, Chula Vista, California
  - Catalina Research Institute, Montclair, California
  - Probe Clinical Research Corporation, Riverside, California
  - Pacific Research Network, San Diego, California
  - Sleep Medicine Specialists of California, San Ramon, California
  - SDS Clinical Trials Inc., Santa Ana, California
  - Provideré Research Inc., West Covina, California
  - Meris Clinical Research, Brandon, Florida
  - Nouvelle Clinical Research, Cutler Bay, Florida
  - Accel Research Sites, DeLand, Florida
  - Research Centers of America, LLC, Hollywood, Florida
  - Canvas Clinical Research, Lake Worth, Florida
  - Florida Lung and Sleep Associates, Lehigh Acres, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - Clinical Site Partners, Miami, Florida
  - Clinical Neuroscience Solutions, Inc - Orlando, Orlando, Florida
  - JSV Clinical Research Study Inc, Tampa, Florida
  - Florida Pediatric Research Institute, Winter Park, Florida
  - Atlanta Center for Medical Research, LLC, Atlanta, Georgia
  - NeuroTrials Research, Atlanta, Georgia
  - Georgia Neurology and Sleep Medicine Assoc, Suwanee, Georgia
  - Javarra Inc-Privia Medical Group, Thomasville, Georgia
  - St. Lukes Clinic - Idaho Pulmonary Associates, Meridian, Idaho
  - Chicago Research Center Inc, Chicago, Illinois
  - OSF HealthCare Saint Francis Medical Center, Peoria, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Centennial Medical Group, Elkridge, Maryland
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Revive Research Institute, Lathrup Village, Michigan
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Neurology Specialists of Monmouth County, West Long Branch, New Jersey
  - Javara Inc - Tryon Medical Partners PLCC, Charlotte, North Carolina
  - Research Carolina Elite, Denver, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Sleep Management Institute (Intrepid), Cincinnati, Ohio
  - UC Health Sleep Medicine, Cincinnati, Ohio
  - University Hospital of Cleveland Medical Center, Cleveland, Ohio
  - Abington Neurological Associate, Abington, Pennsylvania
  - Respiratory Specialists, Wyomissing, Pennsylvania
  - Tribe Clinical Research LL, Greenville, South Carolina
  - OnSite Clinical Solutions LLC/Carolina Cardiology Associates P.A, Rock Hill, South Carolina
  - Chattanooga Research & Medicine, PLLC, Chattanooga, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - The Heights Hospital (HD Heights), Houston, Texas
  - Weill Cornell Medical College, Houston, Texas
  - Lone Star Lung and Sleep Clinic, Houston, Texas
  - Huntsville Research Institute LLC, Huntsville, Texas
  - Epic Medical Research, Red Oak, Texas
  - Element Research Group, San Antonio, Texas
  - South Ogden Family Medicine / CCT Research, South Ogden, Utah
- Canada (8):
  - Canadian Sleep Consultants, Calgary, Alberta
  - Medical Arts Health Research, Kelowna, British Columbia
  - AMNDX, Markham, Ontario
  - West Ottawa Sleep Centre, Ottawa, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Toronto Sleep Institute, Toronto, Ontario
  - Sleep and Alertness Center, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec